CLINICAL TRIAL: NCT02477228
Title: Biliary Cannulation During Endoscopic Retrograde Cholangiopancreatography: Precut Versus Conventional Cannulation. A Prospective Randomized Study
Brief Title: Biliary Cannulation During Endoscopic Retrograde Cholangiopancreatography: Precut Versus Conventional Cannulation
Acronym: ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Gastroenterology surgical center, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Biliary cannulation
Record Dates: First submitted 2015-06-13; First posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Jaundice, Obstructive
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional ERCP (Active Comparator): ERCP was done through the papilla. duration of cannulation, number of trials for cannulation, number of pancreatic cannulation, bleeding during cannulation and its management, need to convert to the other approach in cannulation.
  Interventions: Procedure: conventional ERCP
- Precut ERCP (Active Comparator): ERCP was done through precut from the start duration of cannulation, number of trials for cannulation, number of pancreatic cannulation, bleeding during cannulation and its management, need to convert to the other approach in cannulation.
  Interventions: Procedure: Precut ERCP

INTERVENTIONS:
Procedure: conventional ERCP — ERCP was done through the papilla. duration of cannulation, number of trials for cannulation, number of pancreatic cannulation, bleeding during cannulation and its management, need to convert to the other approach in cannulation.
  Other Names: G1
  Arms: conventional ERCP
Procedure: Precut ERCP — ERCP was done through precut from the start duration of cannulation, number of trials for cannulation, number of pancreatic cannulation, bleeding during cannulation and its management, need to convert to the other approach in cannulation.
  Other Names: G 2
  Arms: Precut ERCP

SUMMARY:
Endoscopic sphincterotomy is now an established method for removal of common bile duct calculi and treatment of papillary stenosis, the sump syndrome and certain cases of ampullary carcinoma. It is also generally performed prior to biliary stent placement .Anatomical variations, papillary stenosis, impacted stones, ampullary tumors, duodenal diverticula, and post-gastrojejunostomy states are some of the reasons behind difficult common bile duct (CBD) cannulations . In these situations, the success of CBD cannulation can be enhanced slightly by using the various accessories designed for this purpose.The aim of this study is to prospectively compare conventional approach and needle knife fistulotomy in cannulation of ampulla of Vater during endoscopic retrograde cholangiopancreatography regarding procedure-related complications as failure of cannulations, bleeding and perforation and postoperative complication

DETAILED DESCRIPTION:
The aim of this study is to prospectively compare conventional approach and needle knife fistulotomy in cannulation of ampulla of Vater during endoscopic retrograde cholangiopancreatography regarding procedure-related complications as failure of cannulations, bleeding and perforation and postoperative complication This a prospective randomized controlled trial comparing two groups of patients who undergo endoscopic retrograde cholangiopancreatography for obstructive jaundice in Gastrointestinal Surgical center, Mansoura University, Egypt. From January 2014 to December 2014.

Group A consists of 50 patients who will undergo conventional approach and group B consists of 50 patients who undergo needle knife fistulotomy for cannulation of the ampulla of Vater. Randomization was done by paramedical personnel in the ERCP unit by taking a number from an envelope.

Data will be registered in a specially prepared sheet for the purpose of the study. Registered data will include: duration of cannulation, number of trials for cannulation, number of pancreatic cannulation, bleeding during cannulation and its management, need to convert to the other approach in cannulation.

Data also included postoperative hospital stay, serum amylase level and postoperative complications as pancreatitis, perforation, bleeding and cholecystitis. Pancreatitis will be also graded according to its severity depending on the duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* all patients (no limit of age) required ERCP calculator and malignant obstructive jaundice

Exclusion Criteria:

* unfit patients history of gastrectomy bleeding tendency larg tumour infiltrating the duodenum

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Successful biliary cannulations | 1 Day
  Successful cannulations of biliary system if the guide wire enter the common bile duct

SECONDARY OUTCOMES:
postprocedure pancreatitis | 30 day
  elevated serum amylase with abdominal pain
postprocedure perforation | 30 day
  duodenal perforation

CONTACTS AND LOCATIONS:
Overall Officials: ayman el nakeeb, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Result] Cortas GA, Mehta SN, Abraham NS, Barkun AN. Selective cannulation of the common bile duct: a prospective randomized trial comparing standard catheters with sphincterotomes. Gastrointest Endosc. 1999 Dec;50(6):775-9. doi: 10.1016/s0016-5107(99)70157-4. PMID 10570335
- [Result] Swan MP, Alexander S, Moss A, Williams SJ, Ruppin D, Hope R, Bourke MJ. Needle knife sphincterotomy does not increase the risk of pancreatitis in patients with difficult biliary cannulation. Clin Gastroenterol Hepatol. 2013 Apr;11(4):430-436.e1. doi: 10.1016/j.cgh.2012.12.017. Epub 2013 Jan 11. PMID 23313840
- [Result] Carr-Locke DL. Biliary access during endoscopic retrograde cholangiopancreatography. Can J Gastroenterol. 2004 Apr;18(4):251-4. doi: 10.1155/2004/364056. PMID 15054501